CLINICAL TRIAL: NCT03261856
Title: Clinical Utility of Carbohydrate Breath Tests in Unexplained GI Symptoms
Brief Title: Clinical Utility of Breath Tests in GI
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Other Study IDs: 1114725
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2018-07

CONDITIONS: Small Intestinal Bacterial Overgrowth; Lactose Intolerance; Fructose Intolerance; Glucose Intolerance
Keywords: Breath test; SIBO; GI
MeSH Terms: conditions — Lactose Intolerance; Fructose Intolerance; Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- small intetsinal bacterial overgrowth: Glucose breath test, 75 g glucose in 250 ml water. Breath samples collected at baseline and every 15 min for 2 hours
- Fructose breath Test: Fructose breath test, 25 g fructose in 250 ml water. Breath samples collected at baseline and every 30 min for 3 hours
- Lactose Breath test: Lactose breath test, 25 g lactose in 250 ml water. Breath samples collected at baseline and every 30 min for 5 hours

SUMMARY:
Bloating, gas, pain and diarrhea are common complaints. Routine investigations are negative; these patients are labeled as IBS. In these patients, whether testing for carbohydrate malabsorption or small intestinal bacterial overgrowth (SIBO) is useful is unclear. Investigators aim to assess the prevalence of SIBO, fructose and lactose intolerance, the usefulness of breath tests, and predictive value of pre-test symptoms.

DETAILED DESCRIPTION:
Abdominal bloating, gas, belching, distension, and diarrhea are common gastrointestinal symptoms that are reported by at least 1/3rd of patients presenting to gastroenterology clinics. When routine endoscopic and radiological tests are negative1, most of these patients are labeled as irritable bowel syndrome (IBS) in gastroenterology practice2. Unfortunately these symptoms persist and these patients remain dissatisfied with their health care and continue to doctor shops or seek remedies from alternative care. Several studies have shown that these symptoms have a significant and negative impact on their quality of life. One possible explanation for their symptom is carbohydrate food intolerance. The Western diet has changed significantly over the last 3 decades. Today, large amounts of fructose are being consumed. This sugar is used as a sweetener in sodas, fruit juices, multiples beverages and candies. Although is naturally present in apples, peaches, pears and oranges, the exponential products and consumption of the synthetic high fructose corn syrup has alarmingly increased fructose consumption. When small amounts are ingested, fructose is completely absorbed from the gut mainly through Glut 5transporter from the intestinal brush border or through facilitated transport along glucose through the Glut 2 transporter5. If a person has either limited absorptive capacity or overwhelms normal absorption capacity by excess ingestion, then malabsorption of fructose ensues. This unabsorbed fructose can serve, as an osmotic load, that draws fluid into the intestinal lumen, causing abdominal bloating, gas, pain and diarrhea 6-7. Likewise lactose is a disaccharide that is present in dairy products and is widely consumed. After ingestion lactose is hydrolyzed in the small intestine by the brush border enzyme lactase into glucose and galactose that are in torn absorbed8. If lactose is malabsorbed by Glut 2, then it will serve as an osmotic load, and get rapidly propelled in to the colon where it is fermented by the colonic bacterial flora, into short chain fatty acid, hydrogen,methane and other gases, this lactose malabsorption produces gas, bloating, flatulence and diarrhea9. About 75% of the world´s population gradually lose their ability to produce the lactase enzyme after age 30 years10-11.

Malabsorption or intolerance of carbohydrates such as fructose and lactose are common and frequently encountered both in the primary care and specialist gastroenterology clinics, but are poorly recognized or treated. Over the last decade, breath testing has emerged as a simple, non invasive method of identifying malabsorption and/ or intolerance to common food ingredients such as fructose12, and lactose13, as well as to identify small intestinal bacterial overgrowth (SIBO)14. However, they are only performed in selected academic centers, and their clinical utility and diagnostic yield largely remains unknown.

Also may the clinical utility of performing a single breath test versus a cumulative battery of breath tests, such as glucose, lactose or fructose breath test, in a patient with unexplained GI symptoms is also not known.

The aims of this study are to investigate a consecutive series of patients with unexplained chronic GI symptoms and examine; 1) the prevalence of SIBO answered by the glucose breath test, fructose and lactose intolerance answered by the fructose y lactose breath test, ; 2) the predictive value of pre-test symptoms in the diagnosis of SIBO or carbohydrate intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Unexplained GI symptoms (gas, bloating, diarrhea, fullness, belching, and abdominal pain)
* Patients who have had normal blood tests and colonoscopy, normal CT or ultrasound scan of the abdomen
* Patients who have completed at least one breath test

Exclusion Criteria:

* Patients with previous GI surgeries (except cholecystectomy, hysterectomy, Nissen funduplication and appendectomy)
* Significant comorbid medical problems (congestive heart failure, chronic renal failure, respiratory failure)
* Cancer
* History of recent antibiotic use (4 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had breath tests as part of routine standard of care to diagnose the unexplained GI symptoms that were abnormal results.
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Actual)
Dates: Start 2011-08-31 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Small Intestinal Bacterial Overgrowth | 3 hour test
  bacterial overgrowth which results in the inability to absorb nutrients
Positive Breath test | 3 hour test
  significant increase in the level of Hydrogen greater than or equal to 20ppm or methane greater than or equal to 15ppm or both above greater than or equal to 15ppm baseline.
Malabsorption | 3 hour test
  significant rise in hydrogen and/or methane levels
Intolerance | 3 hour test
  both the presence of malabsorption and the onset of new symptom or an increase (greater than or equal to 1) in the severity of baseline symptoms
Normal test | 3 hour test
  absence of GI symptoms or change in symptoms during the test together with no significant increase in the levels of hydrogen and methane.
hypersensitivity | 3 hour test
  significant increase (greater than or equal to 1) in the severity of two or more baseline symptoms together with no significant rise in hydrogen or methane levels

CONTACTS AND LOCATIONS:
Overall Officials: Satish SC Rao, MD, PhD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States